CLINICAL TRIAL: NCT04032236
Title: Effect of Oral pH Changes on Smoking Desire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Begum Ergan, Associate Professor, MD, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 437-SBKAEK
Record Dates: First submitted 2019-07-19; First posted 2019-07-25 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Smoking Behaviors
Keywords: caffeine; nicotin; pH
MeSH Terms: conditions — Smoking | interventions — Caffeine; Water

STUDY DESIGN:
Intervention Model Description: case-control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smoking group (Other): 35 smoking case
  Interventions: Other: caffeine
- nonsmoking group (Other): 35 nonsmoking case
  Interventions: Other: caffeine

INTERVENTIONS:
Other: caffeine — At room temperature (18-25 ° C) the same place and standard environment will be done. All involved cases will undergo a dental examination and within 30 minutes three samples of saliva will be taken, including first sample, after coffee drink and after drinking water. The pH of samples will be measured and the smoking cessation rate of the smoking cigarette smoker with simultaneous VAS (VISUAL ANALOG SCALA) will be measured. This data will be compared in-house and non-smoking control group
  Other Names: water

SUMMARY:
Nicotine is a psychoactive substance and its effect is demonstrated by neuronal nicotinic-acetylcholine receptors excreted in the brain and periphery. Psychoactive substances such as nicotine and caffeine play a role in rewarding through the mesolimbic dopaminergic system. The released dopamine produces pharmacological effects that can cause pleasurable emotions. These effects are an important factor in maintaining smoking motivation.

The rate of absorption of nicotine from the buccal mucosa, the rate and amount of dependence, significantly affects the risk. In addition to PH, other factors such as local blood flow, product nematode, size and surface area of the tobacco mixture, constant pH holding capacity, and nicotine content of the tobacco can affect nicotine absorption. To facilitate the absorption of nicotine from the buccal mucosa, various substances that increase absorption have been investigated. Increased alkalinity has been shown to increase nicotine absorption and physiological effects by buffering alkaline pH values with moist snuff products and nicotine gums. Although other factors may affect the nicotine absorption rate in oral tobacco, it is stated that the main factor that determines the rate of nicotine absorption is pH.

Factors that trigger nicotine use include stress in daily life, daily routines, eating and drinking habits, and especially the use of caffeine. The chronic use of caffeine causes tolerance in many of its effects, and the use of nicotine reduces tolerance effects and also potentiates the effects stimulated through the dopaminergic pathway. It has been reported that smokers consume more caffeine than non-smokers.

In the present study, the relationship between oral pH and cigarette demand after caffeine consumption will be investigated. Until now, the relation between cigarette pre- and post-caffeine saliva pH and cigarette smoking has not been investigated. In addition, the effects of drinking behavior and changes in salivary pH on cigarette desire will be investigated and evidence of behavioral methods applied in cigarette smoking cessation treatment will be provided.

DETAILED DESCRIPTION:
Nicotine dependence is accepted as the most common disease and can be treated with medical methods like other diseases. Scientifically proven pharmacotherapy as well as cognitive and behavioral therapy play an important role in reducing cigarette smoking. In this context, it is suggested that the motivation of the person should be questioned, the daily behavioral models should be questioned, the elements triggering the desire for smoking should be identified and the methods of combating them should be developed and the usual vital actions including eating and drinking should be organized. Consumption of acidic foods causes acidic pH in the mouth and salivation increases in order to neutralize it. After meals; tea or coffee, it was reported that smoking desire increases.

Caffeine is another psychostimulant substance found in varying proportions in coffee and tea, and its antagonistic effects on the locomotor system are at adenosine receptors level. Stimulated at low doses and depressed at high doses. Nicotine has a stimulating effect on locomotor activity in chronic use. The chronic use of caffeine causes tolerance in many effects, and nicotine use decreases tolerance effects and also potentiates the effects stimulated through the dopaminergic pathway. It has been reported that smokers consume more caffeine than non-smokers. There are also studies reporting that there is no interaction between caffeine and nicotine and that cocaine consumption increases cigarette smoking as well as epidemiological studies that relate caffeine and nicotine concurrent consumption to pharmacological effects rather than pharmacological effects after food and between studies that are the two most common actions due to stress. However, this effect is not entirely due to the pharmacological effects of caffeine, but influences the intraoral pH and affects the cigarette smoking desire. In this study, the main aim is to investigate the effect of changes in salivary pH on the desire to smoke and how the drinking behavior of water affected this desire.

ELIGIBILITY:
Inclusion Criteria:

1. Not having an active disease
2. Be between the ages of 18 and 45
3. Not using antibiotics in the last two weeks
4. Do not use inhaler treatments
5. Not to have an oral or salivary gland disease
6. One week after menstrual bleeding in female cases
7. At least 10 pack years (P / Y) cigarette story in the case group

Exclusion Criteria:

1. Being an active disease
2. <18 years and> 45 years old
3. Having used antibiotics in the last two weeks
4. Use inhaler treatments
5. Oral and salivary gland disease
6. One week after menstrual bleeding in female cases
7. Being in the luteal phase
8. Menstrual irregularity
9. Being pregnant
10. Taking hormonal treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
To investigate the changes in salivary pH after coffee consumption | 30 minutes after intervention
  salivary pH measurement

SECONDARY OUTCOMES:
to investigate how drinking of water affect the smoking desire | 30 minutes after intervention
  smoking desire will be assessed by visual analog scale with 1 is for minimum and 10 is for maximum desire for smoking

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)